CLINICAL TRIAL: NCT00003254
Title: A Phase II Trial of 5-Fluorouracil Plus 776C85 in Patients With Advanced Resistant Colorectal Cancer
Brief Title: SWOG-S9635 Fluorouracil Plus Ethynyluracil in Advanced Colorectal Cancer Not Responded to Fluorouracil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066138; S9635 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — eniluracil; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 776C85 + 5-FU (Experimental): 776C85, 10mg/m2/dose, PO, Days 1-28 (BID), q 5 wk; 5-FU, 1.0mg/m2/dose, PO, Days 1-28 (BID), q 5 wk.
  Interventions: Drug: ethynyluracil; Drug: fluorouracil

INTERVENTIONS:
Drug: ethynyluracil — 10mg/m2/dose, PO, Days 1-28, q 5wk
  Other Names: 776C85
Drug: fluorouracil — 1.0mg/m2/dose, PO, Days 1-28 BID, q 5wk
  Other Names: 5-FU

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Ethynyluracil may help fluorouracil kill more cancer cells by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of fluorouracil plus ethynyluracil in treating patients with advanced colorectal cancer that has not responded to fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the confirmed response rate to fluorouracil (5-FU) plus ethynyluracil (776C85) in patients with metastatic colorectal cancer that has been demonstrated to be resistant to 5-FU. II. Assess time to progression and survival in this group of patients. III. Assess the frequency and severity of toxicities associated with this treatment.

OUTLINE: Patients are stratified according to relapse while receiving adjuvant therapy (relapse within 12 months of completing adjuvant therapy vs relapse while receiving adjuvant therapy). Patients receive oral doses of ethynyluracil (776C85) and fluorouracil twice daily for 28 days followed by 1 week of rest. Treatment continues every 5 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months the first year, every 4 months the second year, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 35-75 patients will be accrued for this study.

ELIGIBILITY:
* Histologically or cytologically proven metastatic colorectal cancer
* Prior surgery required
* No prior treatment for metastatic disease
* Disease progression while on fluorouracil adjuvant therapy
* Bidimensionally measurable disease
* Age: Over 18
* Performance status: SWOG 0-2
* Hematopoietic: Platelet count at least 100,000/mm3, Absolute granulocyte count at least 1,500/mm3
* Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 3 times ULN (no greater than 5 times ULN if liver involvement)
* Renal: Creatinine clearance at least 50 mL/min
* Other: Must be able to swallow and retain oral medications No nutritional support by gastrostomy feeding tube or parenteral support No intractable vomiting or nausea
* Patients with history of prior malignancy must be currently disease free and off all therapy for that malignancy
* Not pregnant or nursing Fertile patients must use effective contraception
* Biologic therapy: No concurrent immunotherapy Chemotherapy; At least 3 weeks since prior chemotherapy and recovered; No concurrent flucytosine; No other concurrent chemotherapy
* Endocrine therapy: No concurrent hormonal therapy
* Radiotherapy: Prior adjuvant pelvic radiation or radiation to one area of recurrence allowed At least 4 weeks since prior radiotherapy and recovered Total area of bone marrow irradiation must not exceed 25% No concurrent radiotherapy
* Surgery: At least 2 weeks since prior surgery for colorectal cancer and recovered No prior resection of the stomach or small intestine
* Other: No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1998-04; Primary Completion 2002-11 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Confirmed Response Rate | Once every 10 weeks until off treatment
  To assess the confirmed response rate to 5-fluorouracil plus 776C85 in patients with measurable, disseminated colorectal cancer that has been demonstrated to be resistant to 5-fluorouracil.

SECONDARY OUTCOMES:
Progression and Survival | Once every 10 weeks until progression
  To assess time to progression and survival in this group of patients.
Toxicities | Once each week during treatment
  To assess the frequency and severity of toxicities associated with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia G. Leichman, MD, Study Chair — Albany Medical College
Locations (86):
- United States (86):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Leichman CG, Chansky K, Macdonald JS, Doukas MA, Budd GT, Giguere JK, Abbruzzese JL; Southwest Oncology Group. Biochemical modulation of 5-fluorouacil through dihydropyrimidine dehydrogenase inhibition: a Southwest Oncology Group phase II trial of eniluracil and 5-fluorouracil in advanced resistant colorectal cancer. Invest New Drugs. 2002 Nov;20(4):419-24. doi: 10.1023/a:1020662113061. PMID 12448660